CLINICAL TRIAL: NCT04428853
Title: Effects of Iyengar Yoga Therapy in the Management of Stress Urinary Incontinence Among
Brief Title: Effects of Iyengar Yoga Therapy in the Management of Stress Urinary Incontinence Among Young Females
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ziauddin University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: SadiaS
Record Dates: First submitted 2020-06-10; First posted 2020-06-11 (Actual); Last update posted 2022-04-13 (Actual); Status verified 2020-06

CONDITIONS: Stress Urinary Incontinence
MeSH Terms: conditions — Urinary Incontinence, Stress

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- exercise (Experimental): A schedule has designed by the researcher for group yoga therapy of the participant twice a week, each session lasting for 75- minutes for the duration of 8 weeks
  Interventions: Behavioral: iyengar yoga

INTERVENTIONS:
Behavioral: iyengar yoga — different yoga postures including warm up, cool down and meditation that incorporate 75 minutes of training

SUMMARY:
the study is aimed to identify the feasibility, safety, and efficacy of iyengar Yoga therapy in the management of stress urinary incontinence among young female

DETAILED DESCRIPTION:
A total of 44 young female participants will be recruited in this study after signing a written consent. Participants will be attending a 1 hour orientation session prior to yoga therapy providing a general introduction that includes principles, effectiveness and use of props in Iyengar yoga. A schedule will be design by the researcher for group yoga therapy of the participant twice a week, each session lasting for 75- minutes for the duration of 8 weeks by a certified yoga instructor and an assistant. Participants will also instruct to practice yoga at home for 1 additional day per week and to record the dates and duration of practice at home. A manual will be given to the participants with written descriptions in both English and Urdu with pictures portraying each of the key yoga postures performed in the classes. Tips on how to practice each posture safely and comfortably and how to adapt each posture to improve incontinence and pelvic floor function will also be provided in the manual.

Protocols for Yoga Group:

The protocols for Iyengar yoga Therapy will be based on 2 days supervised group yoga classes with an additional 1 day of home yoga performed per week for 8-weeks. Each session will be performed for 75 minutes. This protocol will include 5 phases 1) warm up 2) Pranayamas 3) Active Phase 4) Restorative Phase 5) Meditation.

Warm up:

Warm up will be performed with slow movement combined with breathing for 10 minutes in order to increase core body temperature, lubrication of joint, make connection of mind body spirit and improve blood circulation. Four different postures that will be performed by the participants under the supervision of certified yoga therapist includes cat/cow, wag the tail, thoracic rotation and rock backs. Each posture will be repeated with 5-10 breaths (Miller, 2017).

Pranayamas:

This phase will be consisted of 2 kinds of breathing patterns including Bhramari breathing. This will be performed 5 times with the hold of 10 seconds and Nadi Shodhana breathing. This will be repeated 10 times with the hold of 10 seconds.

Active Phase:

Active phase will be focused on 12 Asanas that are performed in Standing, Sitting and supine positions, directly addressing pelvic floor muscles. In standing postures, Trikonasana, Parsvokonasana, Tadasana, Parsvottasana, Virabhadrasana II, Utkatasana whereas, In Sitting postures, Bharadvajasana, Malasana, Baddha Konasana, and In Supine postures participants will instruct to perform Supta Padagushthasana, Supta Baddha Konasana, Salamba Set Bandhasana.

All of the Asanas will be performed with 5 repetitions. Participants will be maintaining each position for the duration of 15 seconds whereas; intermittent rest of 30 seconds will be given between each yoga posture.

Restorative Phase:

This phase will be focused on postures that rejuvenate the body, mind and spirit while reducing stress and tension of the body. It consists of two postures Viparita Karani Variation and Savasana. Participants must stay in each posture for 4-5 minutes. Meditation:

Meditation guided by breath and mind awareness of the whole body for 10 minutes with calm music.

ELIGIBILITY:
Inclusion Criteria:

* Married Females of age 17-40 year
* Diagnosed Cases of Stress Urinary Incontinence due to pelvic floor muscle weakness

Exclusion Criteria:

* Current Urinary Tract Infection (UTI) or hematuria
* Pregnancy
* On pharmacological treatment of SUI
* Any red flags

Ages: 17 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Gender Based: Yes
Enrollment: 44 (Actual)
Dates: Start 2020-08-15 (Actual); Primary Completion 2021-03-15 (Actual); Study Completion 2021-06-30 (Actual)

PRIMARY OUTCOMES:
pelvic muscle strength (Pre treatment) | baseline
  Perineometer is used to to assess pelvic muscle strength
pelvic muscle strength (Post treatment) | 4th week after intervention
  Perineometer is used to to assess pelvic muscle strength
pelvic muscle strength (Post treatment) | 8th week after intervention
  Perineometer is used to to assess pelvic muscle strength
quantity of urine leakage (Pre treatment) | baseline
  1-hour pad test is used to measure the quantity of urine leakage
quantity of urine leakage (Post treatment) | 4th week after intervention
  1-hour pad test is used to measure the quantity of urine leakage
quantity of urine leakage (Post treatment) | 8th week after intervention
  1-hour pad test is used to measure the quantity of urine leakage
Quality of life (Pre treatment) | baseline
  International Consultation on Incontinence Questionnaire-Urinary Incontinence Short Form (ICIQ-UI SF) is used to assess the quality of life. The total score ranges from 0 to 21, interpretation include; 1 to 5 = Mild, 6 to 12 = moderate, 13 to 18 = severe, 19 to 21 = very severe
Quality of life (Post treatment) | 4th week after intervention
  International Consultation on Incontinence Questionnaire-Urinary Incontinence Short Form (ICIQ-UI SF) is used to assess the quality of life. The total score ranges from 0 to 21, interpretation include; 1 to 5 = Mild, 6 to 12 = moderate, 13 to 18 = severe, 19 to 21 = very severe
Quality of life (Post treatment) | 8th week after intervention
  International Consultation on Incontinence Questionnaire-Urinary Incontinence Short Form (ICIQ-UI SF) is used to assess the quality of life. The total score ranges from 0 to 21, interpretation include; 1 to 5 = Mild, 6 to 12 = moderate, 13 to 18 = severe, 19 to 21 = very severe

CONTACTS AND LOCATIONS:
Overall Officials: sadia shafaq, Principal Investigator — Ziauddin University
Locations (1):
- Ziauddin university, Karachi, Sindh, Pakistan

IPD SHARING:
Plan to Share IPD: No